CLINICAL TRIAL: NCT05596669
Title: Assessment of Analgesic Effect of Ketamine Vs Ketamine Magnesium Infusion and Their Effect on Postoperative Morphine Consumption After Surgical Nephrectomy
Brief Title: Analgesic Effect of Ketamine Vs Ketamine Magnesium Infusion and Their Effect on Postoperative Morphine Consumption
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nirvana Ahmed 02
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Nephrectomy
Keywords: Ketamine; Ketamine Magnesium,; Analgesic,; morphine consumption,; Nephrectomy
MeSH Terms: interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Effect of Ketamine on Postoperative Morphine Consumption (Active Comparator): cases in Group I received infusion of 0.15 mg/kg/h for the duration. Following a parenteral bolus dose of magnesium and ketamine (0.3mg/kg),
  Interventions: Drug: Ketamine
- Effect of Ketamine Magnesium on Postoperative Morphine Consumption (Active Comparator): cases in Group II received Ketamine Magnesium group were given a continuous infusion of (0.15mg/kg/h) of ketamine and (10mg/kg/h) of magnesium
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — to examine the pain-relieving effects of ketamine vs ketamine magnesium infusion, as well as their influence on postoperative morphine consumption following nephrectomy; the secondary goal is to assess hemodynamic effects and pain severity
  Other Names: Ketamine Magnesium; Morphine

SUMMARY:
Ketamine and magnesium-ketamine are two analgesics that are being studied for use as adjuvants. They were shown to have anaesthetic and analgesic properties, and as a consequence of this finding, it has been postulated that they may have a role in minimising the requirement for analgesic drugs during the postoperative period. The major objective of the research was to examine the pain-relieving effects of ketamine vs ketamine magnesium infusion, as well as their influence on postoperative morphine consumption following nephrectomy; the secondary goal is to assess hemodynamic effects and pain severity.

DETAILED DESCRIPTION:
Renal necrosis factor (RN) therapy, which includes ipsilateral adrenalectomy, was first utilized to treat renal cortical tumours in 1969. A radical nephrectomy is a surgical surgery in which the whole kidney, as well as the surrounding fat and, in some cases, the adrenal gland and lymph nodes, are removed. This operation is carried out as an inpatient .

Opioid use, on the other hand, can result in considerable side effects and adverse events, which can result in much longer hospital stays and higher postsurgical hospital costs. Although opioid-based analgesia is essential for postoperative pain management, opioid usage may have serious adverse effects .

Finding techniques to limit opioid intake in the postoperative period is essential because cases that got increased opioid dosages are more likely to have the negative effects. Using non-opioid analgesics alongside opioid analgesics, known as analgesia of multi-modes, to enhance post-operative pain management while reducing the usage of the opioids. .

Ketamine, also and magnesium-ketamine are two analgesics wich are non-opioid that are being studied for use like opioid analgesic adjuvants. They were discovered to have anaesthetic and analgesic properties, and it has been proposed that as a result of this discovery, they may have a great contribution in reducing the need for postoperative analgesic medications .

ELIGIBILITY:
Inclusion Criteria:

* Patients with elective nephrectomy

Exclusion Criteria:

* Pregnant women
* Cases with severe chronic disease as liver cell failures, CHF
* cases with allergies to ketamine and magnesium sulphate
* cases with a history of current regular use of (analgesic, anticonvulsant, antidepressant)
* chronic pain.
* mental illness.

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Measurement of Post-operative Pain | 24-hour analgesic after nephrectomy
  Assessment of the pain post-operatively in patients with pain score as : Total scores vary from 0 to 10 in this method, with a higher score indicating more severe pain,The Ramsay sedation scale was utilized to gauge postoperative sedation levels.

CONTACTS AND LOCATIONS:
Overall Officials: Nirvana Elshalakany, Professor, Principal Investigator — Department of Anesthesia and I.C.U. faculty of Medicine October six university, Egypt
Locations (1):
- October 6 University Hospital, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided